CLINICAL TRIAL: NCT02242864
Title: Micardis® / MicardisPlus® Monitoring of Morning Hypertension and Metabolism II
Brief Title: Study to Evaluate the Effect of the Treatment With Micardis® or MicardisPlus® on Blood Pressure
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.506
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertension and diabetes mellitus
  Interventions: Drug: Micardis®; Drug: MicardisPlus®

INTERVENTIONS:
Drug: Micardis®
Drug: MicardisPlus®

SUMMARY:
The primary objective was to evaluate the effect of the treatment with Micardis® or MicardisPlus® on blood pressure. Secondary objectives were the effect of Micardis® / MicardisPlus® on metabolic parameters (triglycerides, cholesterol, LDL blood glucose, insulin Homeostasis Model Assessment (HOMA)-index and HbA1c) in patients with essential hypertension and diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hypertension
* Diabetes mellitus

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with hypertension and diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in systolic blood pressure (SBP) | Baseline, after 6 months
Change from Baseline in diastolic blood pressure (DBP) | Baseline, after 6 months

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 6-point scale | after 6 months
Assessment of metabolic effect on a 3-point scale | after 6 months
Change from Baseline in laboratory parameters | Baseline, after 6 months
  Metabolic parameters - Triglyceride, total cholesterol, blood glucose, insulin, HOMA-Index, HbA1c
Assessment of tolerability by investigator on a 5-point scale | after 6 months
Number of patients with adverse events | up to 6 months